CLINICAL TRIAL: NCT04541407
Title: A Phase 1 Study of Temozolomide in Combination With Targeted Therapy for NSCLC Patients With CNS Progression on Either Osimertinib or Lorlatinib
Brief Title: Temodar Plus Tyrosine Kinase Inhibitors for Progressive CNS Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-0138.cc; NCI-2020-13878 (Other: CTRP)
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Non Small Cell Lung Cancer; CNS Progression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Temozolomide; osimertinib; lorlatinib

STUDY DESIGN:
Intervention Model Description: This is a phase I, 3 + 3 dose escalation study of Temozolomide plus osimertinib, and temozolomide plus lorlatinib. The two drug combinations will each be examined separately in the 3 + 3 dose escalation schema to determine the MTD(Maximum tolerated dose) and RP2D(Recommended phase 2 dose).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exon 19 deletions or L858R point mutations in exon 21 (Experimental): Will include patients with exon 19 deletions or L858R point mutations in exon 21 of the epidermal growth factor receptor (EGFR) gene. Temozolomide plus Osimertinib will be the study drug combination administered. Osimertinib will be given at a fixed dose of 80 mg daily for dose level 1, with a potential to increase to 160 mg daily for dose level 2. Temozolomide will be started at a dose of 150 mg/m2 on days 1-5 of a 28 day cycle for cycle 1 and if tolerated will be increased to 200 mg/m2 on days 1-5 of a 28 day cycle for cycles 2+. There will be a -1 dose level.
  Interventions: Drug: Temozolomide plus Osimertinib
- Patients with anaplastic lymphoma kinase (ALK) fusions (Experimental): Will include patients with anaplastic lymphoma kinase (ALK) fusions. Temozolomide plus Lorlatinib will be the study drug combination administered. Lorlatinib will be given at a fixed dose of 100 mg daily. Temozolomide will be started at a dose of 150 mg/m2 on days 1-5 of a 28 day cycle for cycle 1 and if tolerated will be increased to 200 mg/m2 on days 1-5 of a 28 day cycle for cycles 2+. There will be a -1 dose level depending on tolerability.
  Interventions: Drug: Temozolomide plus Lorlatinib

INTERVENTIONS:
Drug: Temozolomide plus Osimertinib — Temozolomide is an oral alkylating chemotherapy which has good CNS penetration and has demonstrated CNS responses in both primary brain tumors (e.g., glioblastoma and anaplastic astrocytoma) and in small cell lung cancer (SCLC) brain metastases. Preclinical data from glioblastoma suggests potential synergy of concurrent ALK or EGFR inhibition with temozolomide and early phase trials in glioblastoma are ongoing investigating such combinations. It is felt that combining temozolomide with osimertinib or lorlatinib may be beneficial for patients with progressive CNS disease on either of these TKIs because of the high CNS penetration of temozolomide, good CNS activity of temozolomide in other tumor types and preclinical data from glioblastoma suggesting a potential enhanced effect of concurrent EGFR and ALK/ROS1 inhibition with temozolomide.
  Arms: Exon 19 deletions or L858R point mutations in exon 21
Drug: Temozolomide plus Lorlatinib — Temozolomide is an oral alkylating chemotherapy which has good CNS penetration and has demonstrated CNS responses in both primary brain tumors (e.g., glioblastoma and anaplastic astrocytoma) and in small cell lung cancer (SCLC) brain metastases. Preclinical data from glioblastoma suggests potential synergy of concurrent ALK or EGFR inhibition with temozolomide and early phase trials in glioblastoma are ongoing investigating such combinations. It is felt that combining temozolomide with osimertinib or lorlatinib may be beneficial for patients with progressive CNS disease on either of these TKIs because of the high CNS penetration of temozolomide, good CNS activity of temozolomide in other tumor types and preclinical data from glioblastoma suggesting a potential enhanced effect of concurrent EGFR and ALK/ROS1 inhibition with temozolomide
  Arms: Patients with anaplastic lymphoma kinase (ALK) fusions

SUMMARY:
This trial is testing two novel combinations (temozolomide plus osimertinib OR temozolomide plus lorlatinib) which have not been evaluated in clinical trials. Thus, the exact benefits of these novel combinations are unclear. However, based on the mechanism of action of temozolomide and CNS(Central Nervous System) penetration/activity in other tumor types, it is hypothesized that adding temozolomide to osimertinib or temozolomide to lorlatinib may provide improvement in CNS disease control in patients with CNS progression on either of these latter two TKIs (Tyrosine kinase inhibitors).

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Male or female subject ≥ 18 years old
4. ECOG performance status 0-2
5. Stage IV NSCLC with progression of disease in the CNS on osimertinib 80 mg daily for patients with EGFR activating mutations (EGFR exon 19 deletions or EGFR L858R exon 21 point mutations) -OR- Stage IV NSCLC with progression of disease in the CNS on lorlatinib 100 mg daily for patients with ALK fusions
6. Evaluable CNS disease is required, measurable CNS disease is not required
7. Patients who are on corticosteroids must be on stable or decreasing doses of corticosteroids for at least 14 days.
8. Adequate hematologic function defined as:

   * ANC ≥ 1.5 x 10^9/L
   * Hemoglobin ≥ 9 g/dL
   * Platelets ≥ 150 x 10^9/L
9. Adequate hepatic function defined as:

   * Total bilirubin ≤1.5 x upper limit of normal (ULN). For subjects with Gilbert's Disease, Total bilirubin ≤3 x ULN
   * ALT and AST ≤3 x ULN. For subjects with documented liver metastases, ALT and AST ≤5×ULN
10. Adequate renal function defined as:

    * Estimated glomerular filtration rate (eGFR) ≥ 40 mL/minute as determined using the Cockcroft-Gault formula
11. Patients must be capable of taking oral medication and have no known gastrointestinal malabsorption disorder.
12. Patients must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
13. Brain MRI with contrast is required to have demonstrated progressive CNS disease or an LP with cytology is required to have demonstrated progressive leptomeningeal disease on osimertinib or lorlatinib within 21 days of starting study drugs. CT of brain with contrast can be used to demonstrate progressive disease if patients have a documented anaphylaxis to gadolinium contrast and/or other contraindication to MRI (e.g., severe claustrophobia that cannot be managed with anxiolytics).
14. Patients must not be pregnant. Women/men of reproductive potential must have agreed to use an effective contraceptive method (see section 6.6 for list of effective methods). Women must use an effective contraceptive method during the study and for 6 months following the last dose. Men having sex with women of reproductive potential are required to use effective contraception during the study and for 6 months following the last dose. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" (see section 6.6 for list of effective contraceptive methods) also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a sideeffect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures. Women of reproductive potential are not to be nursing during the study and for six months following the last dose of all study drugs.
15. Women on the lorlatinib arm who are of reproductive potential agree to use a non-hormonal method of contraception during the study and for the time periods outlined above.

Exclusion Criteria:

1. Patients with compound mutations in EGFR will be excluded from this study. Compound mutations are defined as 2 or more mutations in the EGFR tyrosine kinase domain with the following exceptions:

   1. C797S and EGFR exon 19 deletion or EGFR exon 21 point mutation and
   2. T790M mutation and EGFR exon 19 deletion or EGFR exon 21 point mutation.
2. Prior therapy with temozolomide.
3. Patients must not receive surgery or radiation as local therapies for the progressing CNS disease for which they are being enrolled on this trial. Ventriculoperitoneal shunt placement will be allowed for leptomeningeal disease with symptomatic hydrocephalis. Radiation or surgery for progressing extra-CNS disease is allowed.
4. Patients with a history of an allergic/hypersensitivity reaction to any component of temozolomide, dacarbazine, osimertinib (for temozolomide plus osimertinib arm) or lorlatinib (for temozolomide plus lorlatinib arm).
5. Grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., patients with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia.
6. Patients with a history of baseline QTcF interval greater than 470 msec on electrocardiogram for the osimertinib plus temozolomide arm only.
7. Unstable or clinically significant concurrent medical condition, psychiatric illness or social situation that would, in the opinion of the investigator, jeopardize the safety of a subject and/or their compliance with the protocol.
8. Clinically significant acute infection requiring systemic antibacterial, antifungal, or antiviral therapy. Suppressive therapy for chronic infections allowed, for example:

   Subjects with HIV/AIDS with adequate antiviral therapy to control viral load would be allowed. Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy.
9. Treated with any investigational drug or chemotherapy within 3 weeks or ≤ 5 half-lives of first dose of study treatment.
10. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years.
11. Patient is not taking any prohibited medications listed in section 6.4. (Strong CYP3A inducers should be stopped greater than 3 half-lives prior to starting study drugs for patients on either study drug combination. Moderate inducers of CYP3A should be stopped greater than 3 half-lives prior to starting study drugs for patients receiving lorlatinib plus temozolomide. Strong CYP3A inhibitors should be stopped greater than 3 half-lives prior to starting study drugs for patients receiving lorlatinib plus temozolomide.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to 3.5 years
  Adverse events will be determined by the common terminology criteria for adverse events version 5.0

SECONDARY OUTCOMES:
CNS response rate | Up to 3.5 years
  Central Nervous System response rate according to the Response assessment in neuro-oncology (RANO) criteria per investigator assessment. Evaluable CNS lesions may not have been previously irradiated unless they are definitively progressing following radiation and prior to enrollment on the study.
Extra-CNS response rate | Up to 3.5 years
  Extra-CNS response rate according to response evaluation criteria in solid tumors (RECIST) v1.1 per investigator assessment.
Overall response rate | Up to 3.5 years
  Overall response rate including both RANO criteria for CNS response rate and RECIST v1.1 for extra-CNS response rate per investigator assessment.
Incidence of improvement in neurological function | Up to 3.5 years
  Incidence of improvement in neurological function on two successive exams when compared to baseline as determined by one of two study neuro-oncologists
Progression free survival (PFS) | Up to 3.5 years
  PFS will be defined as time from enrollment until development of CNS progressive disease according to the RANO criteria, development of extra-CNS disease progression according to RECIST v1.1 or death.
CNS PFS | Up to 3.5 years
  CNS PFS will be defined as time from enrollment until development of CNS progressive disease per investigator assessment according to the RANO criteria or death.
Extra-CNS PFS | Up to 3.5 years
  Extra-CNS PFS will be defined as time from enrollment until development of progressive disease outside the CNS per investigator assessment according RECIST v1.1 or death.
Overall Survival | Up to 3.5 years
  OS will be defined as time from enrollment until death.Patients alive at date of end of study visit will be censored for survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jose E Pacheco, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No